CLINICAL TRIAL: NCT03125213
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety, Efficacy, and Pharmacokinetics of AL-3778 in Combination With Peginterferon Alpha-2a in Treatment Naïve Chronic Hepatitis B Subjects Who Are HBeAg-positive
Brief Title: A Study Evaluating AL-3778 in Combination With Peginterferon Alpha-2a in Chronic Hepatitis B Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-3778-1003
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peg-IFN plus AL-3778 (Active Comparator)
  Interventions: Drug: AL-3778; Drug: Peginterferon Alfa-2A
- Peg-IFN plus matching placebo (Placebo Comparator)
  Interventions: Drug: Peginterferon Alfa-2A; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: AL-3778 — AL-3778 tablets
  Arms: Peg-IFN plus AL-3778
Drug: Peginterferon Alfa-2A — Peginterferon Alfa-2A for subcutaneous injection
Drug: Placebo Oral Tablet — Placebo to Match AL-3778 tablet
  Arms: Peg-IFN plus matching placebo

SUMMARY:
This is a Phase 2a, multi-center, randomized, double-blind, placebo-controlled study evaluating the safety, efficacy, and pharmacokinetics (PK) of AL-3778 in combination with Peg-IFN in subjects with Hepatitis B e antigen (HBeAg) positive CHB virus infection who are treatment-naïve.

The study will consist of a screening phase , a double-blind treatment phase followed by treatment with Peg-IFN alone, and a post-treatment follow-up phase.

Approximately 30 subjects to complete the study. Eligible subjects will be randomized into 2 treatment arms in a 2:1 ratio (active:placebo) to receive one of the following treatments:

* Arm A: Peg-IFN plus AL-3778 (N=20)
* Arm B: Peg-IFN plus matching placebo (N=10)

ELIGIBILITY:
Inclusion Criteria:

1. A female subject must be of non-childbearing potential
2. Subjects must have CHB infection, documented by serologic profile consistent for CHB infection at screening:

   1. serum HBsAg positive (for >6 months)
   2. serum IgM anti-HBc negative
3. Subjects are treatment-naïve and are serum HBeAg positive with:

   1. serum HBV DNA >=20,000 IU /mL at screening
   2. HBsAg >250 IU/mL at screening
   3. ≥2× upper limit of normal (ULN) ALT and ≤5× ULN at screening

Exclusion Criteria:

1. Positive test for hepatitis A virus immunoglobulin, hepatitis delta antibody (Ab), hepatitis C Ab, human immunodeficiency virus (HIV) Ab and/or evidence of clinically relevant active infection that would interfere with study conduct or its interpretation would also lead to exclusion.
2. Positive test for anti-HBs antibodies and anti-HBe antibodies.
3. Subjects must have low levels of liver fibrosis that is classified as Metavir F0-F2
4. Any history or current evidence of hepatic decompensation
5. Subjects must have absence of hepatocellular carcinoma
6. Subject with evidence of retinopathy on retinal fundus photographs
7. Exclusions related to interferon use for the purposes of this study
8. Subjects with one or more of the following laboratory abnormalities at screening

   1. serum creatinine elevation >1.0× ULN
   2. hemoglobin <11 g/dL [males], <10.5 g/dL [females]
   3. platelet count <125× 109 cells/L
   4. absolute neutrophil count <1.0× 109 cells/L
   5. total bilirubin >1.0× ULN; unless known Gilbert's Disease or Dubin-Johnson Syndrome
9. Subjects having received an investigational agent or investigational vaccine, or having received a biological product within 12 weeks or 5 half-lives (whichever is longer) prior to baseline (first intake of study drugs).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-12 (Estimated); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Mean change (measured in log10 IU/mL) in serum HBsAg from baseline at Week 24. | Day 1 to Week 24

SECONDARY OUTCOMES:
Incidence and severity of AEs | Screening to Week 72
Incidence and severity of laboratory abnormalities | Screening to Week 72
Incidence of serious adverse events (SAEs). | Screening to Week 72
Incidence and severity of AEs leading to study drug discontinuation. | Screening to Week 72
Changes in serum HBV DNA over time | Day 1 to Week 72
Proportion of subjects with ALT normalization | Day 1 to Week 72
Incidence and severity of hepatic flares on treatment | Day 1 to Week 48
Incidence and severity of hepatic flares off-treatment. | Week 48 to week 72
Proportions of subjects with HBeAg loss and/or seroconversion. | Day 1 to Week 72
Proportions of subjects with HBsAg loss and/or seroconversion. | Day 1 to Week 72
Changes in serum HBsAg and serum HBeAg levels over time. | Day 1 to Week 72
Proportion of subjects experiencing a viral breakthrough on treatment. | Day 1 to Week 48
Assess emergence of treatment-associated mutations during study treatment and follow-up with a focus on subjects with treatment failure | Day 1 to Week 72
Individually derived Bayesian estimates of AL-3778 Steady state plasma concentration (C0h) | Week 2
Individually derived Bayesian estimates of AL-3778 area under the plasma concentration curve vs time (AUC0-12h) | Week 2
AL-3778 maximum observed plasma concentration (Cmax) | Week 2
AL-3778 Steady state plasma concentration (C0h) | Week 2
AL-3778 area under the plasma concentration curve vs time (AUC0-12h) | Week 2

CONTACTS AND LOCATIONS:
Overall Officials: William Kennedy, Study Director — Alios Biopharma Inc.

IPD SHARING:
Plan to Share IPD: No